CLINICAL TRIAL: NCT05927831
Title: Comparison of the Effectiveness of Grape Seed Extract (GSE) and Low-level Laser Therapy in the Management of Dentin Hypersensitivity: A Randomized Control Trial
Brief Title: Grape Seed Extract VS Low Level Laser Therapy for Dentin Hypersensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manipal University College Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Anchu Rachel Thomas, Associate Professor Dr., Manipal University College Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 018/2023
Record Dates: First submitted 2023-06-03; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Grape Seed Extract; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Grape seed extract (Experimental): grape seed extract with 95% proanthocyanins will be applied topically to the hypersensitive dentin area for 10 minutes, followed by rinsing with water.
  Interventions: Drug: Grape Seed Extract
- Low-level laser therapy (Experimental): The low-level laser diode treatment of 810 nm will be performed using a commercially available diode laser device. The device will be set at a wavelength of 810 nm, with a power output of 0.5 watts tip of diameter 300 μ in non-contact mode starting at a distance of 5-6 mm away from the hypersensitive tooth area and slowly approaching within a distance of 2-3mm in a scanning motion covering the entire hypersensitive tooth area for a period of 30 seconds to 1 minute.
  Interventions: Device: Low-level laser therapy
- Combination of low-level laser therapy and grape seed extract (Experimental): Grape seed extract will be applied topically to the hypersensitive dentin area for 10 minutes, followed by low-level laser diode treatment.
  Interventions: Drug: Grape Seed Extract; Device: Low-level laser therapy

INTERVENTIONS:
Drug: Grape Seed Extract — Grape seed extract will be applied in the form of a gel on the tooth surface
  Other Names: GSE
  Arms: Combination of low-level laser therapy and grape seed extract; Grape seed extract
Device: Low-level laser therapy — The device will be set at a wavelength of 810 nm, with a power output of 0.5 watts tip of diameter 300 μ in non-contact mode
  Arms: Combination of low-level laser therapy and grape seed extract; Low-level laser therapy

SUMMARY:
Dentin hypersensitivity (DH) is a common clinical problem frequently seen in dental patients. According to Splieth et al., the prevalence of dentin hypersensitivity is 3-98% in adult population.DH is described as a short, sharp pain or discomfort that responses to certain stimuli, typically thermal, tactile, osmotic or chemical, due to exposed dentinal surface which can be explained by the hydrodynamic theory.

The laser is a narrow, focused beam of light emitted to vaporise, fuse, melt, or seal dentinal tubules using laser heat to induce hydroxyapatite crystals for recrystallisation of the mineral component of dentine. The obliteration of dentinal tubules is caused by heat generated by laser beam which inhibits the transmission of the stimulus in the dentinal tubules.

Grape seed extract contains proanthocyanidins (PA) which is able to bind to proline-rich proteins, like collagen, and contributes in enzyme proline hydroxylase activity that is essential for the biosynthesis of collagen in the dentin. The cross-linking action of collagen fibrils in dentin also able to prevent mineral loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least three sensitive tooth by gingival recession or tooth wear >2 scores on the VAS scale.
* Tooth wear index score <3 (Smith and Knight tooth wear index)
* Systemically healthy patient.
* 20-50 years of age.

Exclusion Criteria:

* Teeth with caries, cracked teeth, mobile teeth and pulpitis.
* Deep periodontal pockets (probing depth >6 mm), periodontal surgery within the previous 3 months.
* Recent desensitizing therapy
* systemic diseases and gastric diseases (GERD)
* Allergy to active ingredients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
The patients' dentin hypersensitivity levels will be measured using a visual analogue scale (VAS) | 1st day
  The patients' dentin hypersensitivity levels will be measured using a visual analogue scale (VAS)(0 to 10) before and after treatment.
The patients' dentin hypersensitivity levels will be measured using a visual analogue scale (VAS) | 3rd day
  The patients' dentin hypersensitivity levels will be measured using a visual analogue scale (VAS)(0 to 10) after treatment.
The patients' dentin hypersensitivity levels will be measured using a visual analogue scale (VAS) | 7th day
  The patients' dentin hypersensitivity levels will be measured using a visual analogue scale (VAS)(0 to 10) after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tun Yi Darren Ong, Principal Investigator — Manipal University College Malaysia; Li Jia Ong, Principal Investigator — Manipal University College Malaysia; Ju Wen Lim, Principal Investigator — Manipal University College Malaysia; Wei Nee Lim, Principal Investigator — Manipal University College Malaysia; Gursimrendeep Kaur, Principal Investigator — Manipal University College Malaysia
Locations (1):
- Manipal University College Malaysia, Melaka Tengah, Melaka, Malaysia

IPD SHARING:
Plan to Share IPD: No